CLINICAL TRIAL: NCT03579992
Title: Myoelectric Computer Interface to Reduce Muscle Co-activation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Marc Slutzky, Associate Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00042554
Record Dates: First submitted 2018-06-28; First posted 2018-07-09 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Occupational Therapists were blinded to intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 60-minute Isometric (Experimental): 60-min Isometric MyCI training: EMG-controlled game training for 60-minutes per session
  Interventions: Behavioral: 60-min isometric MyCI training
- 90-minute Isometric (Experimental): 90-min Isometric MyCI training: EMG-controlled game training for 90-minutes per session
  Interventions: Behavioral: 90-min isometric MyCI training
- 90-minute Movement (Experimental): 90-min movement MyCI training: EMG-controlled game training for 90-minutes per session
  Interventions: Behavioral: 90-min movement MyCI training

INTERVENTIONS:
Behavioral: 60-min isometric MyCI training — EMG-controlled in-lab training with arm restrained for 60 minutes per session
  Arms: 60-minute Isometric
Behavioral: 90-min isometric MyCI training — EMG-controlled in-lab training with arm restrained for 90 minutes per session
  Arms: 90-minute Isometric
Behavioral: 90-min movement MyCI training — EMG-controlled in-lab training without restraint for 90 minutes per session
  Arms: 90-minute Movement

SUMMARY:
This study examines whether in-lab training with a myoelectric-computer interface (MyCI) can reduce abnormal muscle co-activation after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors at least 6 months after stroke onset
* Persistent moderate to severe arm impairment
* Increased arm tone

Exclusion Criteria:

* Substantial impairment of vision, memory, language or concentration
* Botulinum toxin use in the affected arm
* Concomitant participation in another research study on the arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity | 6 weeks
  Scale 0-66, total score

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity | 10 weeks
  Scale 0-66, total score
Wolf Motor Function Test | 6 and 10 weeks
  Timed test
Motor Activity Log | 6 and 10 weeks
  30-question test, total score

OTHER OUTCOMES:
Modified Ashworth Scale | 6 and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc Slutzky, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Mugler EM, Tomic G, Singh A, Hameed S, Lindberg EW, Gaide J, Alqadi M, Robinson E, Dalzotto K, Limoli C, Jacobson T, Lee J, Slutzky MW. Myoelectric Computer Interface Training for Reducing Co-Activation and Enhancing Arm Movement in Chronic Stroke Survivors: A Randomized Trial. Neurorehabil Neural Repair. 2019 Apr;33(4):284-295. doi: 10.1177/1545968319834903. Epub 2019 Mar 19. PMID 30888251
- [Derived] Seo G, Kishta A, Mugler E, Slutzky MW, Roh J. Myoelectric interface training enables targeted reduction in abnormal muscle co-activation. J Neuroeng Rehabil. 2022 Jul 1;19(1):67. doi: 10.1186/s12984-022-01045-z. PMID 35778757